CLINICAL TRIAL: NCT06339268
Title: Effects of Preoperative Cognitive and Physical Optimization in the Prevention of Postoperative Cognitive Deficit in Elderly Patients With Lung Resection
Brief Title: Cognitive and Physical Optimization in Prevention of Postoperative Cognitive Deficit in Elderly With Lung Resection
Acronym: COGNITION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Military Medical Academy, Belgrade, Serbia (Other)
Responsible Party: Principal Investigator, Associate Professor Vojislava Neskovic, Associated Professor of Anesthesia and Intensive Care, Military Medical Academy, Belgrade, Serbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MMABelgrade
Record Dates: First submitted 2024-03-11; First posted 2024-04-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Prehabilitation
MeSH Terms: interventions — Cognitive Training; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: After setting the indication for operative treatment, patients who meet the criteria for inclusion in the study, after signing the informed consent, will be randomized into two groups:
  1. The first group (intervention) where the patient will receive preoperative cognitive stimulation and physical therapy for one month before surgical treatment.
  2. The second group (control) where patients receive standard treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients included in the first group will be subjected to psychological testing and preoperative training with the aim of receiving tasks to improve cognitive functions. This technique involves several standardized tests of cognitive stimulation through the Cognifit application on a phone or tablet that patients use three times a week for 20 minutes for a month (from inclusion in the study to scheduled surgery). Also, after consultation with a physiatrist and testing for the presence of weakness syndrome as well as other tests related to the mobility and physical condition of patients, preoperative physical therapy (breathing exercises, walking, climbing stairs) will be carried out in this group of patients. Patients from this group, receive preoperative education on techniques and exercises that they will do immediately postoperatively in bed. Patients will keep a diary of preoperative activities that will be controlled by researchers.
  Interventions: Behavioral: Cognitive training, CogniFit App
- Control group (No Intervention): Patients from the second group will be tested perioperatively with cognitive and weakness syndrome tests and other physiatry tests, but without cognitive intervention and physical therapy, they will be referred for surgery

INTERVENTIONS:
Behavioral: Cognitive training, CogniFit App — A patient will receive preoperative cognitive stimulation and physical therapy for one month before surgical treatment.
  Other Names: Physical therapy
  Arms: Intervention group

SUMMARY:
Postoperative cognitive deficit and its connection with surgery and general anesthesia were first mentioned in the literature in 1955 by Bradford. Cognitive disorders in the postoperative period are postoperative delirium (POD) and postoperative cognitive dysfunction (POCD). POD is an acute dysfunction in cognition, which did not exist preoperatively. Attention deficit disorder is the main symptom of POD and refers to the inability to direct, focus, maintain, or shift attention. Memory impairment, disorientation, or perceptual disturbances may also be present. Cognitive capacity changes in POD patients develop and fluctuate in the first few days after surgery. Unlike POD, there is no formal definition for POCD. Based on data from the existing literature, it is defined as newly diagnosed cognitive deterioration that occurs after surgery. The diagnosis of POCD should be based on pre- and postoperative screening with appropriate psychometric tests. Risk factors for the development of POCD include those related to the surgical procedure, anesthesia, or the patient himself. Compared to less invasive and shorter operations, there is a higher risk of developing POCD after major, invasive, and long-term operations. Additional risk factors are intraoperative (intraoperative bleeding, perioperative transfusion treatment, hypotension) and postoperative complications (respiratory insufficiency, pneumonia, atelectasis, bronchospasm, bronchopleural fistula, and pulmonary edema). Presurgical optimization (Prehabilitation) is a widespread concept that aims to improve the general condition of the patient or optimize comorbidities before major surgery. Prehabilitation is primarily focused on improving physical ability and nutritional status, but it is developing in the direction of a multimodal approach that includes measures to reduce stress and anxiety. Psychological factors are increasingly recognized as an essential element of prehabilitation and are often added to prehabilitation programs.

Older patients, who meet the diagnostic criteria for frailty and are at risk of developing postoperative complications such as cognitive function disorders are increasingly

undergoing lung resection. These complications can affect the outcome and speed of postoperative recovery.

DETAILED DESCRIPTION:
After setting the indication for operative treatment, patients who meet the criteria for inclusion in the study, after signing the informed consent, will be randomized into two groups:

1. The first group (intervention) where the patient will receive preoperative cognitive stimulation and physical therapy for one month before surgical treatment.
2. The second group (control) where patients receive standard treatment. Randomization will be performed using computer randomization by doctors who do not participate in the testing and preoperative preparation of the patient.

Patients included in the first group will be subjected to psychological testing and preoperative training to receive tasks to improve cognitive functions. This technique, known as presurgical cognitive optimization, involves several standardized tests of cognitive stimulation through the cognitive training application (Cognifit) on a phone or tablet that patients use three times a week for 20 minutes for a month (from inclusion in the study to scheduled surgery). Also, after consultation with a physiatrist and testing for the presence of weakness syndrome as well as other tests related to the mobility and physical condition of patients, preoperative physical therapy (breathing exercises, walking, climbing stairs) will be carried out in this group of patients. Patients from this group, in addition to the exercise program they carry out for physical preparation before surgery, receive preoperative education on techniques and exercises that they will do immediately postoperatively in bed. Patients will keep a diary of preoperative activities that will be controlled by researchers.

Patients from the second group will be tested perioperatively with cognitive and weakness syndrome tests and other physiatry tests, but without cognitive intervention and physical therapy, they will be referred for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Older than 60 years
* Elective lung resection operations
* Patients who can use a phone or tablet
* Patients who agreed to participate in the study
* Clinical scale of weakness less than 6
* The American Society of Anesthesiologists (ASA) status I, II, III, IV

Exclusion Criteria:

* Under 60 years of age
* Significant psychiatric comorbidity (schizophrenia, depression, alcoholism)
* Significant neurological comorbidity (dementia, cerebrovascular insult in the last 6 months, parkinsonism)
* Patient's refusal to participate in the study
* The inability of the patient to use a tablet or phone
* The American Society of Anesthesiologists (ASA) status V and VI
* Clinical weakness scale 6 and above

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction | From 1 month preoperatively (schedulling patient for surgery) until 30th postoperative day
  Incidence of newly diagnosed or worsening of the existing postoperative cognitive decline assessed by change in score of MMSE - Mini-Mental State Examination (an 11-question measure that tests five areas of cognitive function: orientation, registration, attention, and calculation, recall, and language). On a scale from 0-30 points:
  ≥ 25 points normal cognitive function 19-24 points minor cognitive dysfunction 10-18 points medium cognitive dysfunction
  ≤ 9 points major cognitive dysfunction In this study change of 3 or more points in MMSE between two tests ( pre and postoperative) or between individual participants will be marked as significant
Perioperative depression and anxiety | From 1 month preoperatively (schedulling patient for surgery) until 30th postoperative day
  Perioperative assessment of depression, anxiety, and stress: DAS - depression and anxiety assessment scale (42-item self-report scale measures the negative emotional states of depression, anxiety, and stress)
  Scoring Guide DASS (42) Scoring Depression Anxiety Stress Normal 0-9 0-7 0-14 Mild 10-13 8-9 15-18 Moderate 14-20 10-14 19-25 Severe 21-27 15-19 26-33 Extremely Severe 28+ 20+ 34+
  Results are assessed between the intervention group and control
Postoperative delirium | First postoperative day
  Incidence of newly diagnosed postoperative delirium: CAM-ICU (Confusion Assessment Method for the ICU) using CAM-ICU Flowsheet:
  Step 1. Acute Change or Fluctuating Course of Mental Status: yes (delirium positive) or no (CAM-ICU negative) Step 2. Inattention: 0 - 2 errors (CAM-ICU negative) or > 2 errors go to next step Step 3. Altered Level of Consciousness (the Richmond Agitation-Sedation Scale - RASS): from -5 (unarousable - no response to voice or physical stimulation) to +4 (combative). Anything other than 0 (alert and calm) goes to the next step.
  Step 4. Disorganized thinking: 0-1 errors (not delirious) or > 1 error (delirious) Feature 1 plus 2 and either 3 or 4 present = CAM-ICU positive
Functional status and postoperative recovery | From 1 month preoperatively (schedulling patient for surgery) until 30th postoperative day
  Assessment of the functional status and speed of recovery - Clinical frailty scale: from 1 (very fit) to 9 (terminally Ill). Only patients marked as less than 6 are included in the study.
  Any change in the assessment score is marked as significant
Functional status and postoperative recovery | From 1 month preoperatively (schedulling patient for surgery) until 30th postoperative day
  Assessment of the functional status and speed of recovery - the New mobility score is a composite score of the patient's ability to perform:
  * indoor walking,
  * outdoor walking
  * shopping
  providing a score between zero and three (0: not at all, 1: with help from another person, 2: with an aid, 3: no difficulty) for each function. The total score can be from 0 to 9, with 9 indicating a high functional level.
Postoperative recovery | From 1st til 5th postoperative day
  Assessment of the speed of recovery - A test of functional recovery: 10 items for assessing basic activities by a six-level ordinal scale 0 (activity not achieved) -5 (fully independent and secure). Total scores can range from 0 to 50 (from inability to perform any activity to complete independence.) Speed of recovery will be assessed with a comparison of the scores during the first 5 postoperative days.
Functional status and postoperative recovery | From 1 month preoperatively (schedulling patient for surgery) until 30th postoperative day
  Assessment of the functional status and speed of recovery Timed up and go test is performed by measuring the time for the following sequence of actions:
  1. Stand up from the chair.
  2. Walk to the line on the floor at a normal pace.
  3. Turn.
  4. Walk back to the chair at a normal pace.
  5. Sit down again.
  Mobility is assessed based on time to complete the test:
  < 10 seconds = normal < 20 seconds = good mobility; can walk outside alone; does not require a walking aid < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid

SECONDARY OUTCOMES:
Overall outcome: Complication rate | From surgery until 30th postoperative day
  Complication rate will be presented as % of patients within the groups who develop:
  * Respiratory failure
  * Pneumonia
  * Atelectasis
  * Bronchospasm
  * Bronchopleural fistula
  * Air leak
  * Pulmonary edema
Overall outcome: Morbidity | From surgery until 30th postoperative day
  Morbidity will be presented as % of patients within the groups who develop any kind of complication or illness postoperatively during the period of follow-up
Overall outcome: Mortality | From surgery until 30th postoperative day
  Mortality will be presented as overall and % of deaths in the study population and both groups

CONTACTS AND LOCATIONS:
Overall Officials: Vojislava Neskovic, PhD, Principal Investigator — Military Medical Academy, Bulgaria
Locations (1):
- Military Medical Academy, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that are collected during the trial, after identification will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] BEDFORD PD. Adverse cerebral effects of anaesthesia on old people. Lancet. 1955 Aug 6;269(6884):259-63. doi: 10.1016/s0140-6736(55)92689-1. No abstract available. PMID 13243706
- [Background] Strom C, Rasmussen LS, Sieber FE. Should general anaesthesia be avoided in the elderly? Anaesthesia. 2014 Jan;69 Suppl 1(Suppl 1):35-44. doi: 10.1111/anae.12493. PMID 24303859
- [Background] Needham MJ, Webb CE, Bryden DC. Postoperative cognitive dysfunction and dementia: what we need to know and do. Br J Anaesth. 2017 Dec 1;119(suppl_1):i115-i125. doi: 10.1093/bja/aex354. PMID 29161395
- [Background] Carli F. Prehabilitation for the Anesthesiologist. Anesthesiology. 2020 Sep;133(3):645-652. doi: 10.1097/ALN.0000000000003331. No abstract available. PMID 32358253
- [Background] Daiello LA, Racine AM, Yun Gou R, Marcantonio ER, Xie Z, Kunze LJ, Vlassakov KV, Inouye SK, Jones RN, Alsop D, Travison T, Arnold S, Cooper Z, Dickerson B, Fong T, Metzger E, Pascual-Leone A, Schmitt EM, Shafi M, Cavallari M, Dai W, Dillon ST, McElhaney J, Guttmann C, Hshieh T, Kuchel G, Libermann T, Ngo L, Press D, Saczynski J, Vasunilashorn S, O'Connor M, Kimchi E, Strauss J, Wong B, Belkin M, Ayres D, Callery M, Pomposelli F, Wright J, Schermerhorn M, Abrantes T, Albuquerque A, Bertrand S, Brown A, Callahan A, D'Aquila M, Dowal S, Fox M, Gallagher J, Anna Gersten R, Hodara A, Helfand B, Inloes J, Kettell J, Kuczmarska A, Nee J, Nemeth E, Ochsner L, Palihnich K, Parisi K, Puelle M, Rastegar S, Vella M, Xu G, Bryan M, Guess J, Enghorn D, Gross A, Gou Y, Habtemariam D, Isaza I, Kosar C, Rockett C, Tommet D, Gruen T, Ross M, Tasker K, Gee J, Kolanowski A, Pisani M, de Rooij S, Rogers S, Studenski S, Stern Y, Whittemore A, Gottlieb G, Orav J, Sperling R; SAGES Study Group*. Postoperative Delirium and Postoperative Cognitive Dysfunction: Overlap and Divergence. Anesthesiology. 2019 Sep;131(3):477-491. doi: 10.1097/ALN.0000000000002729. PMID 31166241
- [Background] Wang W, Wang Y, Wu H, Lei L, Xu S, Shen X, Guo X, Shen R, Xia X, Liu Y, Wang F. Postoperative cognitive dysfunction: current developments in mechanism and prevention. Med Sci Monit. 2014 Oct 12;20:1908-12. doi: 10.12659/MSM.892485. PMID 25306127
- [Background] Sugimoto T, Arai H, Sakurai T. An update on cognitive frailty: Its definition, impact, associated factors and underlying mechanisms, and interventions. Geriatr Gerontol Int. 2022 Feb;22(2):99-109. doi: 10.1111/ggi.14322. Epub 2021 Dec 9. PMID 34882939
- [Background] Gracie TJ, Caufield-Noll C, Wang NY, Sieber FE. The Association of Preoperative Frailty and Postoperative Delirium: A Meta-analysis. Anesth Analg. 2021 Aug 1;133(2):314-323. doi: 10.1213/ANE.0000000000005609. PMID 34257192
- [Background] Durrand J, Singh SJ, Danjoux G. Prehabilitation. Clin Med (Lond). 2019 Nov;19(6):458-464. doi: 10.7861/clinmed.2019-0257. PMID 31732585
- [Derived] Neskovic V, Markovic M, Maric N, Kostic S. Effect of preoperative cognitive and physical optimization in the prevention of postoperative cognitive deficit in elderly patients with lung resection - cognition trial. Trials. 2025 Dec 12. doi: 10.1186/s13063-025-08894-8. Online ahead of print. PMID 41387902